CLINICAL TRIAL: NCT06165575
Title: The Effect of Press Needle in the Combination of Ear and Body Acupuncture Points on Visual Analog Scale in Post-Operative Patients of Open Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Suci Sekarini Martayoga, doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23081272
Record Dates: First submitted 2023-11-01; First posted 2023-12-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Post-operative Pain; Spine, Open
MeSH Terms: conditions — Pain, Postoperative; Spinal Dysraphism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Press needle and medication (Experimental)
  Interventions: Device: Press needle
- Sham press needle and medication (Sham Comparator)
  Interventions: Device: Sham press needle

INTERVENTIONS:
Device: Press needle — Press needle is a very small needles (1-3 mm long) that are 'pressed' onto acupuncture point and are held in place with a small, sterile surgical adhesive patch.
  Arms: Press needle and medication
Device: Sham press needle — Sham press needle is a surgical adhesive patch placed on acupuncture points
  Arms: Sham press needle and medication

SUMMARY:
Postoperative pain is pain that arises after a surgical procedure, resulting from trauma during the surgical incision process. It is generally acute in nature and is accompanied by an inflammatory response. Spinal surgery is a surgical procedure used to address issues typically involving pain in the spinal or back area. Commonly used postoperative analgesics are opioid types administered intravenously. All types of opioids exhibit similar side effects, particularly in terms of respiratory depression, which can lead to hypoxia and respiratory arrest. Other side effects include nausea, vomiting, itching, decreased intestinal motility leading to ileus, and constipation.

The press needle acupuncture, a specialized acupuncture needle developed from intradermal needles, is being used. The advantage of the press needle is its minimally invasive nature, relative affordability, safety, and the ability to continuously stimulate acupuncture points for several days, generally without causing serious side effects.

This study aims to determine the effectiveness of the combined therapy of press needle acupuncture and medication in treating postoperative pain in patients who have undergone open spinal surgery. The study follows a double-blind randomized clinical trial design and is conducted at the inpatient units of Dr. Cipto Mangunkusumo National General Hospital (Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo), University of Indonesia Hospital (Rumah Sakit Universitas Indonesia), and Fatmawati General Hospital. The research is a collaboration between the Medical Acupuncture Department of Faculty of Medicine at the University of Indonesia and the Orthopedics and Traumatology Department. The study employs press needle acupuncture on 8 acupuncture points, 4 ear acupuncture points, and 4 body acupuncture points.

There are three hypothesis for this trial included, first there is a change in the mean pain intensity before the placement of press needles and 24 hours after open spine surgery, following the placement of press needles, in the press needle and medication group at LI4 Hegu, LR3 Taichong, ear acupoint MA TF-1 Shenmen, and MA AT-1 Thalamus compared to the change in mean pain intensity before the placement of sham press needles and 24 hours after open spine surgery, following the placement of sham press needles in the sham press needle and medication group, as measured using the visual analog scale. Second there is a lower mean postoperative pain intensity in the press needle and medication group at LI4 Hegu, LR3 Taichong, ear acupoint MA TF-1 Shenmen, and MA AT-1 Thalamus compared to the sham press needle and medication group, as measured using the visual analog scale at 24 hours and 72 hours after open spine surgery. Third, there is a higher score for postoperative pain management quality in the press needle and medication group at LI4 Hegu, LR3 Taichong, ear point MA TF-1 Shenmen, and MA AT-1 Thalamus compared to the sham press needle and medication group, as assessed using the American Pain Society Patient Outcome Questionnaire Revised questionnaire at 24 hours after open spine surgery

The outcome of this research is the intensity of pain scores measured using the visual analog scale assessed prior to press needle acupuncture insertion, 24 hours post-operation, and 72 hours post-operation. Additionally, the quality of postoperative pain management is assessed using the American Pain Society Patient Outcome Questionnaire Revised (APS-POQ-R) at 24 hours post-operation.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18 years to <= 65 years.
* Patients who have undergone open spine surgery using a conventional method, which involves a surgical procedure with an incision along the spine area for therapeutic purposes, not limited to the entire spine, with or without the use of implants, due to various pathologies other than malignancies.
* Patients are returned to regular inpatient rooms post-surgery.
* Willing to participate in the study until completion.
* Patients with VAS (Visual Analog Scale) >= 6.

Exclusion Criteria:

* Having ear shape abnormalities.
* Wound/infection at acupuncture point areas.
* Having allergies to patches and/or stainless steel.
* Suffering from malignancies.
* Fever > 38°C.
* Taking pre-operative anti-nausea medication.
* Having a history of vertigo complaints

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 24 hours and 72 hours post operative
  The visual analog scale is measured using a visual ruler with a line scale of 10 cm, where patients are asked to draw a line on the ruler according to the pain they are experiencing. Pain scale measurements are taken at 24 hours post-operation and 72 hours post-operation, where a lower scale indicates better progress, which indicates less pain

SECONDARY OUTCOMES:
The American Pain Society Patient Outcome Questionnaire Revised | 24 hours post operative
  The American Pain Society Patient Outcome Questionnaire Revised is a questionnaire designed to assess the quality of postoperative pain management. This questionnaire consists of 6 aspects, pain severity, adverse effects, interference to different activities including sleep, emotional state, perception of care, and nonpharmacological therapies.
  It has 12 items, which rated on 11-point continuous scale from 0 - 10 where 10 signifies the highest score. Frequency of pain and pain relief were measured using worst pain and frequency of pain in 24 h. pain-related interference to activities in bed like turning, repositioning, or out the bed like walking, sitting, standing, and sleep were observed. They were further categorized into: no interference (0), mild (1-3), moderate (4-6), and severe (7-10). Side effect include nausea, drowsiness, itching, dizziness, whereas anxiety, depression, frightened, and helpless behavior were evaluated in emotional state.

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - RSUPN Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region
  - RS Universitas Indonesia, Depok, West Java
  - RSUP Fatmawati, Jakarta

IPD SHARING:
Plan to Share IPD: No